CLINICAL TRIAL: NCT04245592
Title: Fibromyalgia and Oxidative Stress. Influence of the Olive Oil Consumption
Brief Title: Fibromyalgia and Olive Oil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Jaén (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Principal Investigator, Francisco Molina Ortega, Associate professor, University of Jaén
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AGR-6235
Record Dates: First submitted 2020-01-19; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia
Keywords: nutritional intervention; olive oil; nitric oxide; inflammation; cortisol; lipid profile
MeSH Terms: conditions — Fibromyalgia; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients were blinded to the kind of olive oil consumed using unlabeled bottles.
  A coding number in the blood samples of the patients were used to blind the Investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra Virgin Olive Oil (Experimental): Women with fibromyalgia will consume Extra Virgin Olive Oil.
  Interventions: Dietary Supplement: Extra Virgin Olive Oil
- Refined Olive Oil (Experimental): Women with fibromyalgia will consume Refined Olive Oil.
  Interventions: Dietary Supplement: Refined Olive Oil

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil — Before beginning the 3-week dietary trial, participants will conduct a 2-week washout period during which they consumed ROO (50 ml daily for 2 weeks) because they are part of a population that consumes olive oil regularly. After thar, patients of this groups will consume 50 ml/day of organic EVOO for 3 weeks. Biochemical markers and clinical parameters in each participant will be determine before and after the 3-week treatment period.
  Arms: Extra Virgin Olive Oil
Dietary Supplement: Refined Olive Oil — Before beginning the 3-week dietary trial, participants will conduct a 2-week washout period during which they consumed ROO (50 ml daily for 2 weeks) because they are part of a population that consumes olive oil regularly. After thar, patients of this groups will consume 50 ml/day of ROO for 3 weeks. Biochemical markers and clinical parameters in each participant will be determine before and after the 3-week treatment period.
  Arms: Refined Olive Oil

SUMMARY:
We have recently reported a prothrombotic state in patients with fibromyalgia that may increase the risk of thrombosis-related cardiovascular disease in these patients. Several studies have shown the cardioprotective, antithrombotic and antiinflammatory properties of olive oil. The objective of the study is to investigate the effect of consumption of two types of olive oils with different antioxidant content on thrombosis-related parameters, nitric oxide, inflammation, lipid profile and cortisol as well as on health-related parameters in women with fibromyalgia.

DETAILED DESCRIPTION:
Aim:

The goal of the present study is to investigate the effects of two olive oils with different antioxidant content on cardiovascular risk factors (blood-coagulation parameters, platelet indices, red blood cell count, inflammatory markers, lipid profile, nitric oxide and cortisol) in patients diagnosed with fibromyalgia. The investigators will determine thrombosis-related parameters (fibrinogen levels, prothrombin time, prothrombin activity, cephaline time, platelet count, platelet distribution width [PDW], mean platelet volume [MPV], plateletcrit, red blood cell [RBC] count, neutrophil-to-lymphocyte ratio [NLR], and platelet-to-lymphocyte ratio [PLR]), inflammatory markers (interleukin 6 [IL-6], IL-10, C-reactive protein [CRP], erythrocyte sedimentation rate (ESR)), nitric oxide levels, lipid profile, and cortisol levels.

Participants:

This study will be carry out in accordance with the provisions of the Declaration of Helsinki of the World Medical Association.

The research group will contact a Spanish association of patients with fibromyalgia, AFIXA (Association of Fibromyalgia of Jaén, Spain) to find patients to participate in the study. The researchers will convene patients in the laboratory of the Faculty of Health Sciences of the University of Jaén (Spain) to obtain several data of interest (age, BMI, other chronic diseases, pregnancy, lactation and medication). Based on these data, the investigators will select the fibromyalgia group. In a second visit to the laboratory, all patients will sign an informed consent form, the blood samples will be taken and the they will complete several questionnaires (Fibromyalgia Impact Questionnaire, Visual Analogic Scale, Short Form 12 Health Survey).

The women with fibromyalgia will be previously diagnosed with fibromyalgia by a professional rheumatologist and met the American College of Rheumatology (ACR) criteria for fibromyalgia. Exclusion criteria will be the presence of any other chronic disease (diabetes mellitus, hypertension, rheumatoid arthritis, hepatitis, cancer or ischemic heart disease), dyslipidemia, pregnancy, lactation or grade II obesity (BMI ≥ 35 kg/m2). None of the participants will being treated with anticoagulants, corticosteroids, estrogens, analgesics or anti-inflammatory drugs, and will be only included if they had stopped using them at least 2 months before the start of our study. None will consume alcohol regularly, and all will be non-smokers. All the participants will be sedentary.

Study Design: A randomized, controlled, double-blind nutritional trial will carry out. The trial will consist of the consumption of 50 ml/day of one of the two organic olive oils with different antioxidant content, EVOO or ROO, over 3 weeks. A short-term nutritional trial, such as the present one, may offer certain advantages with respect to a long-term trial, as it allows patients to adhere to a stricter and more controlled diet in relation to the intake of other antioxidants. In this way, the possible interference of other antioxidants can be limited, as can interference from possible changes in the lifestyles of the patients, which could also alter the results.

The participants will be randomly assigned to one of the two groups: EVOO and ROO. Before beginning the 3-week dietary trial, participants will conduct a 2-week washout period during which they consumed ROO (50 ml daily for 2 weeks) because they are part of a population that consumes olive oil regularly. Biochemical markers and clinical parameters in each participant will be determine before and after the 3-week treatment period.

Organic olive oils will obtained from Olifarma S.L. (Granada, Spain). The olive oils will be similarly packaged, and participants will be blinded as to the type of olive oil they will consume. Participants will consume the treatment olive oil raw but will use ROO for cooking in order to maintain their ingestion of antioxidants unchanged. The investigators will supply ROO for cooking in sufficient quantity for the whole family. The researchers will estimate the participants' intake by means of a 24-hr recall that they will complete for 3 days (2 working days and a day off) at the beginning of the trial. The investigators will use the average of the values obtained over the 3 days to calculate participants' energy intake (kcals/day) and intake of macronutrients (carbohydrates [g/day], lipids [g/day], and protein [g/day]) and micronutrients, especially those that may have an antioxidant effect, including vitamin C, vitamin A, copper, zinc, and selenium. Based on this analysis, the investigators will provide all participants with dietary recommendations, focusing on the aspects that each should improve. Data of the weight of the participants at the beginning and end of the trial will record. The investigators will request that participants return all the treatment olive oil containers (the consumed and unconsumed containers) at the end of the trial for control of the olive oil consumption (i.e., a count of the empty and full containers each participant will return).

Blood collection and preparation of blood samples: After overnight fasting, venous blood will be taken in the early morning from the antecubital vein into several tubes with anticoagulant and anticoagulant-free tubes. The blood of the anticoagulant-free tubes will be allowed to clot for 30 min at room temperature. The anticoagulant and anticoagulant-free tubes will then be centrifuged at 3500 rpm for 5 min at 4°C to obtain plasma and serum samples, respectively. The blood will be always drawn at the same time of day to avoid circadian variations. Thrombosis-related parameters (fibrinogen levels, prothrombin time, prothrombin activity, cephaline time, platelet count, platelet distribution width [PDW], mean platelet volume [MPV], plateletcrit, red blood cell [RBC] count, neutrophil-to-lymphocyte ratio [NLR], and platelet-to-lymphocyte ratio [PLR]) and erythrocyte sedimentation rate (ESR) were determined in plasma samples. Inflammatory markers (interleukin 6 [IL-6], IL-10, C-reactive protein [CRP]), nitric oxide levels, lipid profile, and cortisol levels were measured in serum samples.

Clinical Characteristics of Participants: The investigators will obtain demographic and clinical data from participants´ interview and questionnaires. The same specialist will carry out all the measurements and tests throughout the study. The questionnaires will be completed immediately after the blood was drawn. The researchers will evaluate functional capacity in daily living activities in patients with fibromyalgia using the Spanish version of the Fibromyalgia Impact Questionnaire (FIQ). The FIQ score, which is the instrument most often used by researchers to estimate fibromyalgia severity, ranges from 0 to 100. Self-reported musculoskeletal pain will be assessed in fibromyalgia patients by a Visual Analogue Scale (VAS; 10 cm). For both of these instruments, higher scores reflect worse symptomatology. The investigators will assess the physical (Physical Component Summary, PCS-12) and mental (Mental Component Summary, MCS-12) health status of patients and controls using the Spanish version of the 12-Item Short-Form Health Survey (SF-12). Scores range from 0 to 100, with lower values reflecting worse health status.

Determination of biochemical parameters

Nitric oxide (NO) Measurement: NO production was indirectly quantified by measuring nitrate/nitrite and S-nitrose compounds (NOx) using an ozone chemiluminescence-based method. The thawed serum aliquots were deproteinized with NaOH 0.8 N and ZnSO4 16% solutions. The total amount of NOx will be determined as previously described (Rus et al., 2011) using the purge system of Sievers Instruments, model NOA 280i (GE Analytical Instruments, Colorado (CO), USA).

Determination of Inflammatory Markers: The IL-6 level will be determined by a chemiluminescent immunoassay using the Access Immunoassay Systems (Beckman Coulter). Levels of IL-10 will be measured by a chemiluminescent immunoenzymatic assay using an MLX™ luminometer (Dynex Technologies, Chantilly, VA). CRP will be measured using an AU 5800 analyzer (Beckman Coulter).

Cortisol Measurement: Cortisol level will be determined in serum samples by a fluorescence polarization immunoassay using an AxSYM analyser (Abbott Laboratories, Illinois (IL), USA).

Determination of Lipid Profile: Serum lipid profile (total cholesterol, high-density lipoprotein [HDL]-cholesterol, triglycerides, apolipoprotein A1, and apolipoprotein B) will be measured by a spectrophotometric procedure using an OLYMPUS AU 5400 analyzer (Beckman Coulter). Low-density lipoprotein (LDL)-cholesterol levels will be estimated indirectly with the Friedewald equation. The level of homocysteine will be determined by a fluorescence polarization immunoassay using an AxSYM analyzer (Abbott Laboratories). The researchers will determine lipid peroxidation by measuring thiobarbituric acid reactive substances (TBARS), which are a good indicator of lipid peroxidation, a major marker of oxidative stress. TBARS will be determined spectrophotometrically in plasma samples following the manufacturer's recommendations (TBARS Assay Kit, OXItek, Catalog. 0801192).

Determination of thrombosis-related parameters: Blood-coagulation parameters (fibrinogen levels, prothrombin time, prothrombin activity and cephaline time) will be determine in plasma samples using the BCS XP analyzer (Siemens Healthineers, Erlangen, Germany). The researchers will measure determinants of platelet function (platelet count, platelet distribution width [PDW], and mean platelet volume [MPV]), and red blood cell (RBC), neutrophil and lymphocyte counts in plasma samples by flow cytometry using the ADVIA 2120 analyzer (Siemens Healthineers, Erlangen, Germany).

Sample size assessment: The sample size has been estimated using the Ene 3.0 software (GlaxoSmithKline). Sample size has been estimated based on the levels of malondialdehyde (Gassió et al., 2008). With an unilateral hypothesis, assuming a probability of type I error of 5%, a β risk of 0.10, with a standard deviation of the effect of 1.4, 10 patients are considered necessary per branch of the study, that is, a total of 20 patients. If 10% of patient losses are assumed, a minimal sample size of 24 patients, 12 for each branch of the study will be needed.

Statistical analysis: The statistical analysis of the data will be performed using the statistical package IBM SPSS Statistics 24 for Windows (SPSS Inc, Chicago, IL). The Kolmogorov-Smirnov test and the Levenne test will be performed to test normality and homoscedasticity, respectively.

To analyze the effect of each olive oil between pre- and post measures, the data that followed a normal distribution and the principle of homoscedasticity of variances were tested by a two-way ANOVA. The statistical significance will be established by applying an unpaired Student's t-test to compare differences between means. Data that did not follow a normal distribution or the principle of homoscedasticity will be tested using the Scheirer-Ray-Hare test, the non-parametric equivalent for two-way ANOVA. The statistical significance will be established by applying the Mann-Whitney U-test to compare differences between means.

To analyze the effect of the type of olive oil, all values will be converted into delta scores (i.e., post-pre values) and thereafter will be tested by unpaired Student's t test or the Mann-Whitney U-test based on normality and homoscedasticity of data.

The effect size will be calculated using the Cohen´s d for parametric tests and the eta squared (η²) for nonparametric tests. Values of Cohen´s d of 0.2, 0.5, and 0.8 correspond to the classical Cohen bands of interpretation of the effect size as small, medium and large, respectively. Values of η² of 0.02, 0.13 and 0.26 correspond to small, medium and large effect size, respectively. The investigators set the level of statistical significance at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women with fibromyalgia will be previously diagnosed with fibromyalgia by a professional rheumatologist and met the American College of Rheumatology (ACR) criteria for fibromyalgia.

Exclusion Criteria:

* Presence of any other chronic disease (diabetes mellitus, hypertension, rheumatoid arthritis, hepatitis, cancer or ischemic heart disease)
* Smokers
* Dyslipidemia
* Pregnancy
* Lactation
* Grade II obesity (BMI ≥ 35 kg/m2)
* Under anticoagulant, corticosteroid, estrogen, analgesic or anti-inflammatory treatment (or they have stopped using them at least 2 months before the start of our study).).
* Patients who consume alcohol regularly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Nitric Oxide | 4 weeks
  NO production will be indirectly quantified by measuring nitrate/nitrite and S-nitrose compounds (NOx) using an ozone chemiluminescence-based method.
Cortisol | 2 weeks
  Cortisol level will be determined in serum samples by a fluorescence polarization immunoassay using an AxSYM analyser
IL-6 | 2 weeks
  Interleukin 6 will be analyzed by chemiluminescent immunoassay using the Access Immunoassay Systems (Beckman Coulter)
Lipid peroxidation | 2 weeks
  Quantitation of thiobarbituric acid reactive substances (TBARS) presence
IL-10 | 2 weeks
  Levels of IL-10 will be measured by a chemiluminescent immunoenzymatic assay using an MLX™ luminometer (Dynex Technologies, Chantilly, VA).
C-Reactive Protein | 2 weeks
  CRP will be measured using an AU 5800 analyzer (Beckman Coulter).
Lipid Profile | 2 weeks
  Serum lipid profile (total cholesterol, high-density lipoprotein [HDL]-cholesterol, triglycerides, apolipoprotein A1, and apolipoprotein B) will be measured by a spectrophotometric procedure using an OLYMPUS AU 5400 analyzer (Beckman Coulter). Low-density lipoprotein (LDL)-cholesterol levels will be estimated indirectly with the Friedewald equation. The level of homocysteine will be determined by a fluorescence polarization immunoassay using an AxSYM analyzer (Abbott Laboratories)
Fibrinogen | 2 weeks
  Will be determined in plasma samples using the BCS XP analyzer (Siemens Healthineers, Erlangen, Germany).
Prothrombin activity | 2 weeks
  Will be determined in plasma samples using the BCS XP analyzer (Siemens Healthineers, Erlangen, Germany).
Cephaline time | 2 weeks
  Will be determined in plasma samples using the BCS XP analyzer (Siemens Healthineers, Erlangen, Germany).
Platelet count | 2 weeks
  Will be measured in plasma samples by flow cytometry using the ADVIA 2120 analyzer (Siemens Healthineers, Erlangen, Germany).
Platelet distribution width [PDW] | 2 weeks
  Will be measured in plasma samples by flow cytometry using the ADVIA 2120 analyzer (Siemens Healthineers, Erlangen, Germany).
Mean platelet volume [MPV] | 2 weeks
  Will be measured in plasma samples by flow cytometry using the ADVIA 2120 analyzer (Siemens Healthineers, Erlangen, Germany).
Red blood cell (RBC) | 2 weeks
  Will be measured in plasma samples by flow cytometry using the ADVIA 2120 analyzer (Siemens Healthineers, Erlangen, Germany).
Neutrophil count | 2 weeks
  Will be measured in plasma samples by flow cytometry using the ADVIA 2120 analyzer (Siemens Healthineers, Erlangen, Germany).
Lymphocyte counts | 2 weeks
  Will be measured in plasma samples by flow cytometry using the ADVIA 2120 analyzer (Siemens Healthineers, Erlangen, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: María Luisa Del Moral, MD, Principal Investigator — University of Jaen
Locations (1):
- Francisco Molina Ortega, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gassio R, Artuch R, Vilaseca MA, Fuste E, Colome R, Campistol J. Cognitive functions and the antioxidant system in phenylketonuric patients. Neuropsychology. 2008 Jul;22(4):426-31. doi: 10.1037/0894-4105.22.4.426. PMID 18590354
- [Background] Rus A, Peinado MA, Blanco S, Del Moral ML. Is endothelial-nitric-oxide-synthase-derived nitric oxide involved in cardiac hypoxia/reoxygenation-related damage? J Biosci. 2011 Mar;36(1):69-78. doi: 10.1007/s12038-011-9006-4. PMID 21451249